CLINICAL TRIAL: NCT05464043
Title: Screening for Diabetes and Pre-diabetes in a Cohort of Pediatric Patients Who Have Received a Liver or Kidney Transplant (DIAB-GRAFT)
Brief Title: Hyperglycemia and (Pre)Diabetes in Pediatric Renal and Liver Transplantation.
Acronym: DIAB-GRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DIAB-GRAFT
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diabetic cohort (Experimental): Patients who receive liver or kidney transplants and immunosuppressive drugs with diabetogenic risk.
  After 14 days of immunosuppressive therapy, all admitted patients will be evaluated for first-line glucose homeostasis. This patient cohort will be referred to as the "diabetes risk cohort".
  Subjects will then be stratified into two groups of patients: those who have developed glycemic dysregulation or diabetes during immunosuppressive therapy, the "diabetic cohort", and those who have not developed glycemic dysregulation or diabetes, the "control cohort". Only those who have developed glycemic dysregulation or diabetes during immunosuppressive therapy, i.e. the "diabetic cohort", will be analysed in more detail with the evaluation of second-line glucose homeostasis at three different times.
  Interventions: Diagnostic Test: evaluation of second line glucose homeostasis

INTERVENTIONS:
Diagnostic Test: evaluation of second line glucose homeostasis — blood samples, urine samples, genetic test, peptide C stimulation test, OGTT, continuous glucose monitoring and questionnaires

SUMMARY:
Background: Diabetes is a common complication of transplantation and is associated with unfavorable medical outcome and increased cardiovascular disease at long term. However, prediabetes defined by an impaired glucose tolerance and/or impaired fasting glucose is rarely sought in pediatric liver (LT) and renal (RT) transplantation, while its presence indicates a high risk of overt diabetes and complications thereof. Early detection of hyperglycemia might mitigate those risks. The objectives of the DIABGRAFT study were to retrospectively (rDIABGRAFT) and longitudinally (pDIABGRAFT) characterize hyperglycemia and (pre)diabetes in a cohort of children with RT or/and LT.

Methods: The investigators retrospectively collected data about 195 children with LT from 2012 and 2019 and twenty children with RT from 2005 to 2019 in Cliniques universitaires Saint Luc to determine the incidence, risk factors and time at onset of chronic hyperglycemia. In addition, the investigators prospectively followed four LT and four RT children between 2019 and 2022 to evaluate the evolution of their glucose metabolism.

DETAILED DESCRIPTION:
BACKGROUND/AIM: Solid organ transplantation (SOT) is therapeutic choice for patient in end-stage renal or liver disease. After transplant, immunosuppressive therapy is necessary to avoid rejection and their use has enabled SOT and considerably improved graft survival and quality of life. However, they are also associated with side effects, including glycemic abnormalities. Most complications observed with immunosuppressants are the presence of hyperglycemia which in the long term may increase the probabilities to develop persistent diabetes. Diabetes affects an ill-defined proportion of transplanted patients (2 to 53%) and in the context of adult liver and renal transplant, it is nonetheless common, and represents approximately 20%. However, the incidence of transient hyperglycemia and the probabilities to develop overt diabetes in pediatric liver and renal transplantation remains unknow, while it is known that both is associated with an unfavorable prognosis (i.e., mortality, graft rejection, increased hospital stay) and an increased cardiovascular event in the long term. Moreover, associated risk factors such as obesity, metabolic syndrome, sedentary lifestyle, or even older age are well known for adult transplant but do not make sense for children transplanted at a very young age. In addition, the use of a non-relevant measure such as fasting blood glucose and a late-onset diabetes marker like HbA1C levels do not allow the early detection of impaired glucose tolerance (IGT) a signal alarm of a prediabetes state. Prediabetes is considered as an intermediate state between normal glucose homeostasis and overt diabetes and represents a major health problem because it is estimated in 2015 that 70% of the prediabetic American citizens (33,5%) will develop diabetes in the period. However, it is rarely sought in pediatric transplantation while the early detection and correction of hyperglycemia was shown to significantly decrease both cardiovascular and diabetes risk. It is therefore essential to develop knowledge on the evolution of glucose dysregulation after a renal and liver transplantation with the implementation of other markers of hyperglycemia or IGT. Then the purpose of the DIABGRAFT study was to assess the incidence and associated risk factors of developing hyperglycemia in renal and liver transplanted children to anticipate it and analyze their glycemic profile during the most critical moment to characterize hyperglycemia, IGT and diabetes.

METHODS: In collaboration with the Pediatric Gastroenterology and Specialized Pediatrics Services (Endocrinology and Nephrology Units) of Cliniques universitaires Saint Luc (CUSL) in Belgium (Brussels), this clinical study will be organized as a retrospective and a prospective trial.

The study included liver and renal transplanted pediatric patients (<18 years of age) at CUSL. Were excluded patients with a history of diabetes (i.e., type 1, type 2, neonatal or monogenic), pancreatitis, Down Syndrome, cystic fibrosis, another transplantation (cardiac, renal) only for liver transplanted patients, patients deceased shortly after transplantation, and patients with incomplete medical record.

Its retrospective part (rDIABGRAFT) consisted of collecting data of pediatric patients who benefited from a liver transplant performed at CUSL between April 2012 and April 2019, or that benefited from a renal transplant in our center between April 2005 and April 2019.

The prospective part (pDIABGRAFT) of the study consisted of a longitudinal glycemic evaluation of renal and liver transplanted children in CUSL between 2020 and 2022 with the use of dynamic endocrine testing. Informed consents were collected from parents and from all children over six years of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone liver and/or kidney transplantation and immunosuppressive treatments such as glucocorticoids, cyclosporin A, tacrolimus and sirolimus, treated and monitored in the gastroenterology and pediatric hepatology department and in the pediatric nephrology department (hospitalized patients and outpatient clinics) of Cliniques universitaires Saint-Luc.
* Informed consent obtained prior to any activity related to the trial. Test activities are all procedures performed as part of the test, including activities to determine test suitability.
* Age of the patient at presentation: 2 years - 18 years.
* For inclusion in the diabetogenic risk cohort: patients under diabetogenic treatment protocols such as glucocorticoids, cyclosporin A and tacrolimus.
* For inclusion in the diabetic cohort: patients under diabetogenic treatment protocols such as glucocorticoids, cyclosporin A and tacrolimus and diabetes diagnosis according to the 2014 guidelines of the International Paediatric and Adolescent Diabetes Society (ISPAD).

Exclusion Criteria:

Diagnosis of type 1 or monogenic diabetes; Palliative care patients; History of pancreatitis (acute or chronic);

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Retrospective study: characterization of hyperglycemia and diabetes after liver or kidney transplantation | Before transplantation until the end of the study (April 2022)
  Incidence and risk factors of hyperglycemia and diabetes after liver or kidney transplantation

SECONDARY OUTCOMES:
Prospective: analysis of impaired glucose tolerance (prediabetes) and diabetes after liver or kidney transplantation | At day 14 post transplantation until 1 month for liver transplant and 9 months for kidney transplant
  Composite of tests and analysis to evaluate glucose homeostasis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lysy, MD, Phd, Principal Investigator — Cliniques Universitaires Saint-Luc UCLouvain
Locations (1):
- Cliniques Universitaires Saint-Luc - UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welsch S, Mailleux V, le Hardy de Beaulieu P, Ranguelov N, Godefroid N, Robert A, Stephenne X, Scheers I, Reding R, Sokal EM, Lysy PA. Characterization, evolution and risk factors of diabetes and prediabetes in a pediatric cohort of renal and liver transplant recipients. Front Pediatr. 2023 Feb 7;11:1080905. doi: 10.3389/fped.2023.1080905. eCollection 2023. PMID 36824650